CLINICAL TRIAL: NCT00305747
Title: Phase I Study of Bioresponse-dim in Non-Metastatic, Hormone-Refractory Prostate Cancer Patients With Rising Serum PSA
Brief Title: Diindolylmethane in Treating Patients With Nonmetastatic Prostate Cancer That Has Not Responded To Previous Hormone Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elisabeth Heath, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000462637; P30CA022453 (NIH); WSU-D-2979; WSU-0507002581
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; adenocarcinoma of the prostate; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BR-DIM (Experimental): BR-DIM will be administered at a starting dose of 75 mg po twice daily. Patients will be instructed to take tablets twice daily with 8 ozs. of water, with/without food. A study calendar will be provided and patients will be asked to fill the appropriate boxes when they take their study capsules. One treatment cycle is 28 days.
  Interventions: Drug: BR-DIM

INTERVENTIONS:
Drug: BR-DIM — 75 mg orally (po) twice daily. May continue treatment for 12 months, however patients will be taken off study if their disease progresses, or have intolerable side effects.
  Other Names: oral microencapsulated diindolylmethane

SUMMARY:
RATIONALE: Diindolylmethane may slow the growth of prostate cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of diindolylmethane in treating patients with nonmetastatic prostate cancer that has not responded to previous hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Establish the maximum tolerated dose, dose-limiting toxicity, and a recommended phase II dose of absorption-enhanced diindolylmethane (BioResponse-DIM^® [BR-DIM]) in patients with nonmetastatic, hormone-refractory prostate cancer and rising serum prostate-specific antigen (PSA) levels.
* Evaluate the toxicities of BR-DIM.

Secondary

* Evaluate the plasma pharmacokinetics of twice daily oral administration of BR-DIM in this patient population.
* Evaluate the effect of BR-DIM supplementation on serum PSA level.
* Correlate changes in expression levels of lymphocytes NF-kB with serum PSA levels in patients taking BR-DIM supplementation.
* Determine quality of life measures in patients taking BR-DIM supplementation.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive oral absorption-enhanced absorption-enhanced diindolylmethane (BioResponse-DIM^® [BR-DIM]) twice daily on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of BR-DIM until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

Quality of life is assessed at baseline, on day 1 of each course, and at the completion of study therapy.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven adenocarcinoma of the prostate
* Prostate specific antigen (PSA)-only failure after local therapy (surgery, radiation therapy, brachytherapy, or cryotherapy)
* Rising PSA despite androgen-deprivation therapy with castrate levels of testosterone (< 50 ng/dL)

  * Two successive rising PSA levels at least 1 week apart
  * PSA ≥ 5 ng/mL
* Patients with a history of combined hormonal therapy must continue luteinizing-hormone releasing-hormone agonist treatment but must demonstrate rising PSA after anti-androgen withdrawal
* No evidence of distant metastasis by bone scan and CT scan
* No known brain metastases requiring active therapy

PATIENT CHARACTERISTICS:

* ECOG performance status ≤ 3
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT and/or SGPT ≤ 2.5 times ULN AND alkaline phosphatase normal OR alkaline phosphatase ≤ 4 times ULN AND SGOT and/or SGPT normal
* Creatinine clearance ≥ 60 mL/min OR creatinine normal
* Fertile patients must use effective contraception
* None of the following conditions within the past 6 months:

  * Myocardial infarction
  * Severe or unstable angina
  * Symptomatic congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Coronary/peripheral artery bypass grafting
* No other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would preclude study participation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 28 days since prior radiotherapy
* At least 28 days since prior investigational agents for treatment of prostate cancer
* At least 4 weeks since prior flutamide
* At least 6 weeks since prior bicalutamide
* No other concurrent antineoplastic agents
* No concurrent warfarin-related anticoagulants
* No concurrent proton-pump inhibitor drugs for gastroesophageal reflux disease (e.g., rabeprazole, esomeprazole magnesium, lansoprazole, omeprazole, or pantoprazole sodium)
* No concurrent micronutrient supplements or dietary soy products

  * One daily multivitamin allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD), Dose limiting toxicity (DLT) & toxicities during study and for 30 days after | During study and for 30 days after

SECONDARY OUTCOMES:
Plasma pharmacokinetics as measured by occurrences of toxicity | At baseline; Cycle 1 Day 1 at 20, 60, 120, 180, 240, and 480 minutes
Serum prostate specific antigen as measured by complete plasma concentration-time profile | At baseline, Day 1 of each cycle and at study termination
Correlate changes in expression levels of NF-kB lymphocytes in with serum prostate specific antigen levels by serum prostate specific antigen level | At baseline, Cycle 2 and study termination
Quality of life (QOL) by Life Orient. Test-Rev., Duke-UNC Func. Social Support Questionnaire, EORTC QOL questionnaire, QLQ-PR25 questionnaire, and the Hosp. Anxiety & Depression Scale | At baseline, day 1 of each cycle and study termination

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth I. Heath, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Detroit, Michigan